CLINICAL TRIAL: NCT03449901
Title: A Phase II Trial of ADI-PEG 20 in Combination With Gemcitabine and Docetaxel for the Treatment of Soft Tissue Sarcoma Osteosarcoma, Ewing's Sarcoma, and Small Cell Lung Cancer
Brief Title: ADI-PEG 20 in Combination With Gemcitabine and Docetaxel for the Treatment of Soft Tissue Sarcoma, Osteosarcoma, Ewing's Sarcoma, and Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201912062-1001; 1R01CA227115-01A1 (NIH)
Record Dates: First submitted 2018-02-20; First posted 2018-02-28 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — ADI PEG20; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: ADI-PEG 20 + Gemcitabine + Docetaxel (Experimental): * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 600 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
  Interventions: Drug: pegylated arginine deiminase; Drug: Gemcitabine; Drug: Docetaxel; Procedure: Tumor biopsy; Procedure: Research blood draw
- Cohort 2: ADI-PEG 20 + Gemcitabine + Docetaxel (Experimental): * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 600 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
  Interventions: Drug: pegylated arginine deiminase; Drug: Gemcitabine; Drug: Docetaxel; Procedure: Tumor biopsy; Procedure: Research blood draw

INTERVENTIONS:
Drug: pegylated arginine deiminase — -Arginine deiminase (ADI) is a recombinant protein cloned from M. hominis, produced in E. coli, and conjugated with PEG of 20,000 mw using a succinimidyl succinate linker. Thus ADI-PEG 20 is an arginine degrading enzyme, ADI, coupled to PEG.
  Other Names: ADI-PEG 20
Drug: Gemcitabine — -Gemcitabine is a nucleoside metabolic inhibitor that exhibits antitumor activity.
  Other Names: Gemzar
Drug: Docetaxel — -Docetaxel is an antineoplastic agent belonging to the taxoid family. It is prepared by semisynthesis beginning with a precursor extracted from the renewable needle biomass of yew plants.
  Other Names: Taxotere
Procedure: Tumor biopsy — * Up to 21 days prior to initiation of ADI-PEG 20 Day -1 (+/- 1 day as long as performed prior to initiation of gemcitabine.
  * Tumor biopsies are mandatory for the first 20 patients amendable to biopsy enrolled at Washington University only (completed as of 05/14/2019) and for all patients enrolled to the SCLC cohort
Procedure: Research blood draw — -Day -7 (pre-treatment), Day -1, and Days 1 and 8 of each cycle

SUMMARY:
The investigators have recently demonstrated that argininosuccinate synthase 1 (ASS1) expression is silenced in 88% of all sarcomas (n=708), and that this loss is associated with a decreased overall survival. Using the extracellular arginine depleting enzyme PEGylated arginine deiminase (ADI-PEG20), an extracellular arginine depleting enzyme, the investigators demonstrated ADI-PEG20 induces a prosurvival metabolic reprogramming in ASS1-deficient sarcomas that redirects glucose into the serine/folate pathway directing the carbons from glucose into pyrimidine biosynthesis, thus sensitizing cells to death by the pyrimidine antimetabolite gemcitabine by using metabolomics. The synthetic lethality was increased by the addition of docetaxel. Therefore a phase II clinical trial of ADI with gemcitabine and docetaxel, a standard second line therapy for soft tissue sarcoma will be conducted to determine if the clinical benefit rate of gemcitabine and docetaxel is improved by the metabolic changes induced by ADI-PEG20.

Recently published data shows that priming ASS1-deficient tumors with ADI-PEG 20 and docetaxel improves the effect of gemcitabine. Therefore, a cohort of patients consisting of ten patients diagnosed with either osteosarcoma or Ewing's sarcoma (ideally five of each), and five patients diagnosed with small cell lung cancer will be included as an exploratory cohort. Enrollment to Cohort 2 will occur concurrently with Cohort 1.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Histologically or cytologically confirmed grade 2 or 3 soft tissue sarcoma that is unresectable or metastatic that would be standardly treated with gemcitabine or gemcitabine and docetaxel. For all others, please contact the principal investigator. Prior surgery for primary or metastatic disease after chemotherapy following a response is allowed.
* Cohort 2: Histologically or cytologically confirmed osteosarcoma, Ewing's sarcoma, or small cell lung cancer that is unresectable or metastatic that have either failed standard of care therapy or would be standardly treated with gemcitabine or gemcitabine and docetaxel.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Treated with at least one line of systemic therapy. The allowable window between treatments is 21 days for chemotherapy or a TKI, or 5 ½ half-lives for a TKI (whichever is shorter), 21 days and progression by CT for immunotherapy, 21 days for RT, 21 days for surgery, or 28 days for an investigational agent.
* Cohort 1: At least 16 years of age.
* Cohort 2: Patients with osteosarcoma or Ewing's sarcoma must be at least 10 years of age. Patients with small cell lung cancer must be at least 18 years of age.
* Cohort 2 (SCLC group ONLY): Must be amenable to biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 2 x institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3 x IULN (or ≤ 5 x IULN if liver metastases are present)
  * Creatinine ≤ 1.5 x IULN OR
  * Creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
  * Serum uric acid ≤ 8 mg/dL (with or without medication control)
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* A history of other high grade malignancy ≤ 5 years previous. Exceptions include basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix, or other tumors discussed with the study PI
* Currently receiving any other investigational agents.
* Prior treatment with ADI-PEG 20, gemcitabine, or docetaxel. Patients treated > one year ago in the adjuvant/neoadjuvant setting with gemcitabine or docetaxel would be allowed to be enrolled on the trial.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial (except for patients with SCLC, see below) because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with SCLC are allowed to enroll with brain metastases provided they are stable and they are at least 3 months post-treatment for brain metastases.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to ADI-PEG 20, gemcitabine, pegylated compounds, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of seizure disorder not related to underlying cancer.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with the study treatment. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mia Weiss, M.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Stanford Medicine, Palo Alto, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient was enrolled, but never initiated treatment.
Groups:
- Cohort 1: ADI-PEG 20 + Gemcitabine + Docetaxel: Patients enrolling to Cohort 1 must be diagnosed with soft tissue sarcoma.
  * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 600 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
- Cohort 2: ADI-PEG 20 + Gemcitabine + Docetaxel: Patients enrolling to Cohort 2 must be diagnosed with osteosarcoma, Ewing's sarcoma, or small cell lung cancer.
  * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 600 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
Period: Overall Study
Arm/Group | Cohort 1: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 2: ADI-PEG 20 + Gemcitabine + Docetaxel
Started | 82 | 15
Completed | 1 (1 patient completed treatment per protocol.) | 0
Not Completed | 81 | 15
Not completed — Progression | 57 | 12
Not completed — Adverse Event | 3 | 0
Not completed — Death | 6 | 2
Not completed — Withdrawal by Subject | 12 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Patient elected for surgical intervention | 1 | 0
Not completed — Patient off for other complicating disease | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 2: ADI-PEG 20 + Gemcitabine + Docetaxel | Total
Number analyzed (Participants) | 82 | 15 | 97
Age, Continuous [Median (Full Range); unit: years] | 57 [16 to 86] | 30 [12 to 71] | 55 [12 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 7 | 52
  Male | 37 | 8 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 78 | 13 | 91
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 71 | 11 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 82 | 15 | 97

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) (Cohort 1 Only)
Description: * PFS: defined as time on study to time patients progressed on the drug combination or death or latest follow-up if progression/death is not observed yet
  * Progressive disease: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Through completion of follow-up (median follow-up 494 days, full range of 5-1500 days).
Population: PFS was evaluated only for Cohort 1; therefore, no participants in Cohort 2 were analyzed for this outcome measure. 2 participants in Cohort 1 were not evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 2: ADI-PEG 20 + Gemcitabine + Docetaxel
Number analyzed (Participants) | 80 | 0
months | 5.0597 [2.9898 to 7.5238] |

2. Secondary Outcome: Overall Survival (OS) (Cohort 1 Only)
Description: -OS: defined as time on study to time of death due to any reasons or latest follow-up (whichever is earlier)
Time Frame: Through completion of follow-up (median follow-up 494 days, full range of 5-1500 days).
Population: OS was evaluated only for Cohort 1; therefore, no participants in Cohort 2 were analyzed for this outcome measure. 7 participants in Cohort 1 were not evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 2: ADI-PEG 20 + Gemcitabine + Docetaxel
Number analyzed (Participants) | 75 | 0
months | 18.1359 [14.0290 to 25.1011] |

3. Secondary Outcome: Clinical Benefit Rate (CBR) (Cohort 1 Only)
Description: * CBR = proportion of patients who have experienced complete response (CR)+ partial response (PR) + stable disease (SD) lasting 24 weeks or longer
  * CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  * PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Through completion of treatment (median treatment of 9 months)
Population: CBR was evaluated only for Cohort 1; therefore, no participants in Cohort 2 were analyzed for this outcome measure. 8 participants in Cohort 1 were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 2: ADI-PEG 20 + Gemcitabine + Docetaxel
Number analyzed (Participants) | 74 | 0
Participants | 27 |

4. Secondary Outcome: Safety and Tolerability of Regimen as Measured by Number and Grade of Adverse Events
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Time Frame: From start of treatment through 30 days after completion of treatment (median treatment of 9 months + 1 month follow-up)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel; Cohort 2, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel: * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 600 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
- Cohort 1, 750 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel: * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 750 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
- Cohort 1, 900 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel: * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 900 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
Arm/Group | Cohort 1, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 1, 750 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 1, 900 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 2, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel
Number analyzed (Participants) | 33 | 25 | 24 | 15
Participants
  Grade 1-2 anemia | 11 | 9 | 12 | 9
  Grade 3-5 anemia | 19 | 11 | 12 | 4
  Grade 3-5 febrile neutropenia | 2 | 3 | 1 | 1
  Grade 1-2 eosiniphilia | 0 | 0 | 0 | 1
  Grade 3-5 mitral valve disease | 1 | 0 | 0 | 0
  Grade 1-2 atrial fibrillation | 0 | 1 | 0 | 0
  Grade 3-5 atrial fibrillation | 0 | 1 | 1 | 0
  Grade 1-2 palpitations | 2 | 0 | 0 | 0
  Grade 3-5 pericardial effusion | 1 | 0 | 0 | 0
  Grade 1-2 sinus bradycardia | 0 | 1 | 0 | 0
  Grade 1-2 sinus tachycardia | 1 | 2 | 0 | 1
  Grade 3-5 sinus tachycardia | 1 | 0 | 0 | 0
  Grade 1-2 chest pain - cardiac | 0 | 0 | 1 | 0
  Grade 1-2 ear pain | 1 | 0 | 0 | 0
  Grade 1-2 vertigo | 1 | 0 | 2 | 0
  Grade 3-5 tinnitus | 0 | 1 | 0 | 0
  Grade 1-2 hyperthyroidism | 0 | 1 | 0 | 0
  Grade 1-2 cataract | 1 | 1 | 0 | 0
  Grade 1-2 blurred vision | 0 | 1 | 0 | 0
  Grade 1-2 watering eyes | 1 | 2 | 2 | 0
  Grade 1-2 retinal tear | 0 | 1 | 0 | 0
  Grade 1-2 dry eye | 0 | 0 | 1 | 0
  Grade 1-2 abdominal distension | 0 | 1 | 0 | 0
  Grade 1-2 abdominal pain | 3 | 1 | 2 | 1
  Grade 3-5 abdominal pain | 0 | 0 | 1 | 0
  Grade 1-2 anal hemorrhage | 0 | 0 | 1 | 0
  Grade 1-2 anal mucositis | 0 | 0 | 1 | 0
  Grade 1-2 ascites | 0 | 0 | 1 | 0
  Grade 3-5 ascites | 0 | 0 | 1 | 0
  Grade 1-2 bloating | 0 | 1 | 0 | 0
  Grade 1-2 colitis | 0 | 1 | 1 | 0
  Grade 1-2 colonic hemorrhage | 0 | 0 | 1 | 0
  Grade 3-5 colonic perforation | 0 | 0 | 1 | 0
  Grade 1-2 constipation | 8 | 5 | 8 | 2
  Grade 1-2 dental caries | 3 | 0 | 0 | 0
  Grade 3-5 dental caries | 1 | 0 | 0 | 0
  Grade 1-2 diarrhea | 10 | 7 | 7 | 1
  Grade 3-5 diarrhea | 0 | 1 | 2 | 1
  Grade 1-2 dry mouth | 1 | 1 | 0 | 0
  Grade 1-2 dyspepsia | 4 | 2 | 3 | 2
  Grade 1-2 dysphagia | 1 | 1 | 0 | 1
  Grade 1-2 fecal incontinence | 0 | 0 | 0 | 1
  Grade 1-2 flatulence | 0 | 0 | 1 | 0
  Grade 1-2 gastroesophageal reflux disease | 1 | 0 | 0 | 1
  Grade 1-2 hematochezia | 1 | 1 | 0 | 0
  Grade 3-5 generalized GI bleed | 0 | 0 | 1 | 0
  Grade 1-2 tooth extraction | 1 | 0 | 0 | 0
  Grade 1-2 hemorrhoids | 0 | 2 | 1 | 0
  Grade 3-5 lower gastrointestinal hemorrhage | 0 | 1 | 0 | 0
  Grade 1-2 lip pain | 1 | 0 | 0 | 0
  Grade 1-2 mucositis oral | 6 | 5 | 3 | 2
  Grade 1-2 nausea | 13 | 8 | 14 | 2
  Grade 1-2 oral pain | 0 | 1 | 0 | 0
  Grade 1-2 rectal hemorrhage | 0 | 1 | 0 | 0
  Grade 3-5 small intestinal obstruction | 2 | 2 | 0 | 0
  Grade 3-5 typhlitis | 0 | 0 | 1 | 0
  Grade 3-5 upper gastrointestinal hemorrhage | 0 | 1 | 0 | 0
  Grade 1-2 vomiting | 6 | 4 | 3 | 4
  Grade 3-5 vomiting | 1 | 0 | 0 | 0
  Grade 1-2 chills | 0 | 1 | 0 | 0
  Grade 5 death NOS | 0 | 0 | 0 | 1
  Grade 1-2 edema face | 0 | 1 | 0 | 0
  Grade 1-2 edema limbs | 9 | 5 | 10 | 2
  Grade 3-5 edema limbs | 1 | 1 | 1 | 0
  Grade 1-2 edema trunk | 0 | 1 | 0 | 0
  Grade 3-5 edema trunk | 0 | 0 | 1 | 0
  Grade 1-2 facial pain | 1 | 0 | 0 | 0
  Grade 1-2 fatigue | 16 | 15 | 10 | 5
  Grade 3-5 fatigue | 7 | 7 | 8 | 0
  Grade 1-2 fever | 5 | 9 | 5 | 1
  Grade 1-2 flu-like symptoms | 1 | 1 | 1 | 0
  Grade 1-2 generalized edema | 5 | 0 | 0 | 0
  Grade 1-2 infusion related reaction | 1 | 0 | 0 | 1
  Grade 1-2 injection site reaction | 3 | 3 | 1 | 1
  Grade 1-2 localized edema | 0 | 0 | 1 | 0
  Grade 1-2 malaise | 0 | 0 | 1 | 0
  Grade 1-2 non-cardiac chest pain | 0 | 1 | 1 | 1
  Grade 3-5 non-cardiac chest pain | 1 | 0 | 1 | 0
  Grade 1-2 pain at injection site | 0 | 2 | 0 | 0
  Grade 1-2 pain | 0 | 0 | 0 | 1
  Grade 3-5 hepatic hemorrhage | 0 | 0 | 1 | 0
  Grade 1-2 allergic reaction | 3 | 0 | 0 | 0
  Grade 3-5 allergic reaction | 1 | 0 | 0 | 0
  Grade 3-5 Celiac disease | 0 | 1 | 0 | 0
  Grade 1-2 bladder infection | 0 | 0 | 1 | 0
  Grade 1-2 bronchial infection | 1 | 0 | 1 | 0
  Grade 1-2 enterocolitis infectious | 1 | 0 | 1 | 0
  Grade 3-5 enterocolitis infectious | 1 | 1 | 0 | 1
  Grade 1-2 eye infection | 1 | 0 | 0 | 0
  Grade 1-2 folliculitis | 1 | 0 | 0 | 0
  Grade 1-2 gum infection | 1 | 0 | 0 | 0
  Grade 3-5 influenza A infection | 1 | 0 | 0 | 0
  Grade 1-2 lung infection | 2 | 1 | 0 | 0
  Grade 3-5 lung infection | 1 | 1 | 2 | 1
  Grade 1-2 papulopustular rash | 1 | 0 | 0 | 0
  Grade 1-2 paronychia | 0 | 0 | 1 | 0
  Grade 3-5 pleural infection | 0 | 0 | 0 | 1
  Grade 3-5 sepsis | 1 | 3 | 4 | 1
  Grade 1-2 sinusitis | 3 | 2 | 0 | 0
  Grade 1-2 skin infection | 0 | 1 | 1 | 0
  Grade 3-5 skin infection | 1 | 0 | 2 | 1
  Grade 1-2 thrush | 3 | 1 | 1 | 0
  Grade 1-2 tooth infection | 1 | 0 | 0 | 0
  Grade 1-2 upper respiratory infection | 2 | 5 | 4 | 0
  Grade 3-5 upper respiratory infection | 1 | 0 | 0 | 0
  Grade 1-2 urinary tract infection | 1 | 0 | 4 | 0
  Grade 3-5 urinary tract infection | 0 | 3 | 1 | 0
  Grade 3-5 wound infection | 0 | 0 | 1 | 0
  Grade 1-2 ankle fracture | 0 | 1 | 0 | 0
  Grade 1-2 bruising | 1 | 0 | 1 | 0
  Grade 1-2 fall | 2 | 1 | 1 | 0
  Grade 3-5 fall | 0 | 1 | 0 | 0
  Grade 1-2 fracture | 2 | 0 | 0 | 0
  Grade 1-2 twisted knee | 1 | 0 | 0 | 0
  Grade 3-5 ileal bleed due to tumor invasion | 1 | 0 | 0 | 0
  Grade 3-5 postoperative hemorrhage | 1 | 0 | 0 | 0
  Grade 1-2 spinal fracture | 0 | 0 | 1 | 0
  Grade 3-5 wound complication | 0 | 0 | 1 | 0
  Grade 1-2 activated partial thromboplastin time prolonged | 1 | 2 | 3 | 0
  Grade 3-5 activated partial thromboplastin time prolonged | 1 | 0 | 2 | 0
  Grade 1-2 alanine aminotransferase increased | 12 | 13 | 8 | 4
  Grade 3-5 alanine aminotransferase increased | 2 | 1 | 3 | 0
  Grade 1-2 alkaline phosphatase increased | 12 | 11 | 13 | 5
  Grade 3-5 alkaline phosphatase increased | 1 | 1 | 0 | 1
  Grade 1-2 aspartate aminotransferase increased | 1 | 7 | 8 | 2
  Grade 3-5 aspartate aminotransferase increased | 0 | 1 | 2 | 0
  Grade 1-2 blood bilirubin increased | 2 | 6 | 6 | 1
  Grade 3-5 blood bilirubin increased | 0 | 0 | 1 | 1
  Grade 1-2 lactate dehydrogenase increased | 2 | 0 | 1 | 0
  Grade 1-2 cardiac troponin I increased | 1 | 1 | 0 | 0
  Grade 3-5 cardiac troponin I increased | 0 | 1 | 1 | 0
  Grade 1-2 cardiac troponin T increased | 0 | 0 | 1 | 0
  Grade 1-2 creatinine increased | 6 | 5 | 9 | 0
  Grade 3-5 creatinine increased | 1 | 0 | 0 | 1
  Grade 1-2 electrocardiogram QT corrected interval prolonged | 1 | 0 | 0 | 0
  Grade 3-5 electrocardiogram QT corrected interval prolonged | 0 | 1 | 0 | 0
  Grade 1-2 INR increased | 4 | 3 | 9 | 0
  Grade 3-5 GGT increased | 0 | 0 | 0 | 1
  Grade 3-5 INR increased | 0 | 1 | 3 | 0
  Grade 3-5 ammonia increased | 0 | 0 | 0 | 1
  Grade 1-2 lipase increased | 0 | 0 | 1 | 0
  Grade 3-5 lipase increased | 0 | 0 | 1 | 0
  Grade 1-2 lymphocyte count decreased | 6 | 7 | 4 | 2
  Grade 3-5 lymphocyte count decreased | 18 | 11 | 20 | 8
  Grade 1-2 neutrophil count decreased | 6 | 1 | 6 | 3
  Grade 3-5 neutrophil count decreased | 19 | 18 | 11 | 7
  Grade 1-2 platelet count decreased | 6 | 5 | 9 | 4
  Grade 3-5 platelet count decreased | 23 | 18 | 12 | 7
  Grade 1-2 weight loss | 0 | 3 | 0 | 2
  Grade 1-2 white blood cell count decreased | 6 | 5 | 5 | 2
  Grade 3-5 white blood cell count decreased | 19 | 17 | 15 | 9
  Grade 3-5 acidosis | 0 | 0 | 1 | 0
  Grade 1-2 anorexia | 5 | 5 | 5 | 2
  Grade 3-5 anorexia | 0 | 1 | 1 | 0
  Grade 1-2 dehydration | 1 | 4 | 1 | 0
  Grade 3-5 dehydration | 0 | 1 | 1 | 0
  Grade 1-2 hypercalcemia | 1 | 2 | 1 | 1
  Grade 1-2 hyperglycemia | 6 | 4 | 5 | 2
  Grade 3-5 hyperglycemia | 0 | 1 | 2 | 0
  Grade 1-2 hyperkalemia | 1 | 1 | 0 | 2
  Grade 3-5 hyperkalemia | 0 | 0 | 1 | 0
  Grade 1-2 hyperlipidemia | 0 | 0 | 1 | 0
  Grade 1-2 hypermagnesemia | 0 | 0 | 1 | 0
  Grade 3-5 hypermagnesemia | 0 | 0 | 1 | 1
  Grade 1-2 hypernatremia | 1 | 1 | 1 | 1
  Grade 1-2 hyperuricemia | 6 | 5 | 6 | 2
  Grade 3-5 hyperuricemia | 2 | 0 | 4 | 0
  Grade 1-2 hypoalbuminemia | 14 | 6 | 13 | 1
  Grade 3-5 hypoalbuminemia | 1 | 2 | 2 | 2
  Grade 1-2 hypocalcemia | 12 | 6 | 11 | 2
  Grade 3-5 hypocalcemia | 3 | 1 | 1 | 2
  Grade 1-2 hypoglycemia | 1 | 1 | 2 | 0
  Grade 3-5 hypoglycemia | 0 | 0 | 2 | 0
  Grade 1-2 hypokalemia | 5 | 6 | 7 | 2
  Grade 3-5 hypokalemia | 2 | 1 | 3 | 1
  Grade 1-2 hyponatremia | 14 | 7 | 11 | 5
  Grade 3-5 hyponatremia | 0 | 0 | 1 | 1
  Grade 1-2 hypophosphatemia | 6 | 1 | 4 | 3
  Grade 3-5 hypophosphatemia | 0 | 3 | 2 | 0
  Grade 1-2 arthralgia | 3 | 3 | 2 | 0
  Grade 1-2 back pain | 4 | 3 | 4 | 0
  Grade 3-5 back pain | 0 | 1 | 1 | 0
  Grade 1-2 bone pain | 3 | 2 | 3 | 2
  Grade 1-2 flank pain | 1 | 1 | 0 | 0
  Grade 1-2 generalized muscle weakness | 4 | 3 | 4 | 1
  Grade 1-2 joint effusion | 0 | 0 | 1 | 0
  Grade 1-2 muscle cramp | 6 | 2 | 0 | 0
  Grade 1-2 muscle weakness lower limb | 0 | 1 | 0 | 0
  Grade 1-2 myalgia | 5 | 7 | 2 | 1
  Grade 1-2 neck pain | 0 | 1 | 0 | 0
  Grade 1-2 pain in extremity | 3 | 2 | 1 | 1
  Grade 1-2 palpable lump RUE | 1 | 0 | 0 | 0
  Grade 1-2 skin pailloma, R hallux | 1 | 0 | 0 | 0
  Grade 3-5 disease progression | 2 | 0 | 2 | 0
  Grade 1-2 tumor pain | 9 | 3 | 0 | 1
  Grade 3-5 tumor pain | 0 | 0 | 0 | 1
  Grade 1-2 concentration impairment | 1 | 1 | 0 | 0
  Grade 1-2 dizziness | 1 | 5 | 2 | 0
  Grade 1-2 dysgeusia | 8 | 5 | 8 | 0
  Grade 1-2 extrapyramidal disorder | 1 | 0 | 0 | 1
  Grade 1-2 headache | 5 | 5 | 3 | 1
  Grade 1-2 plantar sensitivity | 0 | 1 | 0 | 0
  Grade 3-5 cerebral hemorrhage | 0 | 1 | 0 | 0
  Grade 1-2 neuralgia | 1 | 1 | 2 | 0
  Grade 1-2 paresthesia | 2 | 2 | 0 | 0
  Grade 1-2 paresthesia (face) | 0 | 0 | 0 | 1
  Grade 1-2 peripheral sensory neuropathy | 9 | 5 | 10 | 0
  Grade 1-2 phantom pain | 0 | 0 | 1 | 0
  Grade 1-2 presyncope | 2 | 0 | 2 | 0
  Grade 3-5 spinal cord compression | 0 | 1 | 0 | 0
  Grade 3-5 syncope | 2 | 1 | 0 | 0
  Grade 1-2 tremor | 0 | 0 | 1 | 0
  Grade 3-5 agitation | 1 | 0 | 0 | 0
  Grade 1-2 anxiety | 3 | 2 | 0 | 0
  Grade 1-2 confusion | 2 | 2 | 0 | 1
  Grade 3-5 confusion | 1 | 0 | 0 | 0
  Grade 1-2 depression | 4 | 1 | 0 | 1
  Grade 3-5 depression | 1 | 0 | 0 | 0
  Grade 1-2 insomnia | 2 | 3 | 2 | 1
  Grade 1-2 irritability | 0 | 0 | 0 | 1
  Grade 1-2 acute kidney injury | 0 | 1 | 0 | 0
  Grade 3-5 acute kidney injury | 2 | 0 | 1 | 0
  Grade 1-2 dysuria | 1 | 2 | 0 | 0
  Grade 1-2 hematuria | 9 | 3 | 8 | 0
  Grade 1-2 proteinuria | 7 | 7 | 7 | 0
  Grade 1-2 renal calculi | 0 | 1 | 0 | 0
  Grade 1-2 urinary frequency | 0 | 1 | 0 | 0
  Grade 1-2 urinary incontinence | 0 | 1 | 0 | 0
  Grade 1-2 urinary retention | 1 | 1 | 0 | 0
  Grade 3-5 urinary tract obstruction | 1 | 0 | 1 | 0
  Grade 1-2 genital edema | 0 | 0 | 1 | 0
  Grade 1-2 pelvic pain | 0 | 0 | 1 | 0
  Grade 1-2 groin pain | 1 | 0 | 0 | 0
  Grade 1-2 vaginal hemorrhage | 0 | 1 | 0 | 0
  Grade 1-2 allergic rhinitis | 1 | 2 | 0 | 0
  Grade 3-5 bronchial obstruction | 0 | 1 | 0 | 0
  Grade 1-2 cough | 5 | 6 | 5 | 2
  Grade 1-2 dyspnea | 12 | 4 | 6 | 3
  Grade 3-5 dyspnea | 3 | 1 | 1 | 0
  Grade 1-2 epistaxis | 6 | 6 | 3 | 3
  Grade 1-2 hoarseness | 1 | 1 | 1 | 0
  Grade 1-2 hypoxia | 1 | 0 | 0 | 0
  Grade 3-5 hypoxia | 0 | 1 | 1 | 0
  Grade 1-2 laryngeal hemorrhage | 1 | 1 | 0 | 0
  Grade 1-2 laryngeal inflammation | 1 | 1 | 0 | 0
  Grade 1-2 nasal congestion | 1 | 0 | 0 | 0
  Grade 1-2 pleural effusion | 3 | 1 | 2 | 2
  Grade 3-5 pleural effusion | 2 | 0 | 1 | 1
  Grade 3-5 pneumonitis | 1 | 0 | 0 | 0
  Grade 1-2 pneumothorax | 0 | 0 | 0 | 1
  Grade 3-5 pneumothorax | 0 | 0 | 2 | 0
  Grade 1-2 postnasal drip | 0 | 0 | 1 | 0
  Grade 1-2 productive cough | 2 | 2 | 1 | 0
  Grade 3-5 pulmonary edema | 1 | 1 | 0 | 0
  Grade 3-5 respiratory failure | 0 | 1 | 0 | 0
  Grade 1-2 chest pressure with exertion | 1 | 0 | 0 | 0
  Grade 1-2 rhinorrhea | 2 | 2 | 0 | 0
  Grade 1-2 sore throat | 1 | 3 | 1 | 1
  Grade 1-2 wheezing | 1 | 1 | 1 | 0
  Grade 1-2 alopecia | 2 | 2 | 1 | 1
  Grade 1-2 bullous dermatitis | 1 | 0 | 1 | 0
  Grade 1-2 dry skin | 0 | 1 | 0 | 0
  Grade 1-2 hyperhidrosis | 0 | 1 | 1 | 0
  Grade 1-2 nail changes | 0 | 1 | 4 | 0
  Grade 1-2 nail discoloration | 1 | 0 | 0 | 0
  Grade 1-2 nail loss | 1 | 0 | 1 | 0
  Grade 1-2 palmar-plantar erythrodysesthesia syndrome | 0 | 1 | 1 | 0
  Grade 1-2 pruritus | 1 | 1 | 1 | 0
  Grade 3-5 pruritus | 0 | 1 | 0 | 0
  Grade 1-2 rash acneiform | 1 | 0 | 2 | 0
  Grade 1-2 rash maculo-papular | 2 | 1 | 1 | 4
  Grade 3-5 rash maculo-papular | 0 | 1 | 0 | 0
  Grade 1-2 skin atrophy | 1 | 0 | 0 | 0
  Grade 1-2 rash NOS | 1 | 0 | 0 | 0
  Grade 3-5 petechial rash | 0 | 0 | 0 | 1
  Grade 1-2 skin ulceration | 1 | 0 | 0 | 1
  Grade 1-2 urticaria | 1 | 0 | 0 | 0
  Grade 1-2 minor gum transplant | 2 | 0 | 0 | 0
  Grade 1-2 hot flashes | 1 | 0 | 0 | 0
  Grade 1-2 hypertension | 3 | 2 | 0 | 0
  Grade 3-5 hypertension | 1 | 1 | 2 | 0
  Grade 1-2 hypotension | 1 | 3 | 3 | 0
  Grade 3-5 hypotension | 0 | 1 | 0 | 0
  Grade 1-2 lymphedema | 1 | 0 | 0 | 0
  Grade 1-2 thromboembolic event | 0 | 2 | 1 | 0
  Grade 3-5 thromboembolic event | 1 | 1 | 1 | 0
  Grade 1-2 peripheral edema | 0 | 1 | 0 | 0
  Grade 1-2 muscle "tightness" | 1 | 0 | 0 | 0
  Grade 1-2 left hand pain | 1 | 0 | 0 | 0
  Grade 1-2 right axillary pain | 0 | 1 | 0 | 0
  Grade 1-2 right neck stiffness | 0 | 1 | 0 | 0
  Grade 1-2 "frozen thumb" | 0 | 1 | 0 | 0
  Grade 1-2 hip pain | 0 | 0 | 1 | 1
  Grade 1-2 ankle sprain | 1 | 0 | 0 | 0
  Grade 1-2 port site bleed | 0 | 1 | 0 | 0
  Grade 1-2 vaginal cyst | 0 | 1 | 0 | 0
  Grade 1-2 rash NOS on neck | 0 | 1 | 0 | 0
  Grade 1-2 rash NOS on bilateral UE | 0 | 1 | 0 | 0
  Grade 1-2 nail bed pain | 1 | 0 | 0 | 0
  Grade 1-2 feet peeling | 0 | 1 | 0 | 0
  Grade 3-5 leukemia secondary to oncology chemotherapy | 0 | 1 | 0 | 0

5. Secondary Outcome: Number of Participants With Cancer-related Mortality (Cohort 1 Only)
Time Frame: Through completion of follow-up (median follow-up 494 days, full range of 5-1500 days).
Population: Cancer-related mortality was evaluated only for Cohort 1; therefore, no participants in Cohort 2 were analyzed for this outcome measure. 7 participants in Cohort 1 were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 2: ADI-PEG 20 + Gemcitabine + Docetaxel
Number analyzed (Participants) | 75 | 0
Participants | 47 |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment through 30 days after the completion of study treatment. The range of collection was 35 to 870 days, with a median following time of 87 days. All-cause mortality was collected from start of treatment through completion of follow-up. The range of collection was 5 to 1500 days, with a median follow-up time of 494 days.
Groups:
- Cohort 1, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel: Patients enrolling to Cohort 1 must be diagnosed with soft tissue sarcoma.
  * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 600 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
- Cohort 1, 750 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel: Patients enrolling to Cohort 1 must be diagnosed with soft tissue sarcoma.
  * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 750 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
- Cohort 1, 900 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel: Patients enrolling to Cohort 1 must be diagnosed with soft tissue sarcoma.
  * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 900 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
- Cohort 2, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel: Patients enrolling to Cohort 2 must be diagnosed with osteosarcoma, Ewing's sarcoma, or small cell lung cancer.
  * ADI-PEG 20 will be given on Day -7 of Cycle 1 and then on Days 1, 8, and 15 of each subsequent cycle. Cycles are 21 days. ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m2 via intramuscular injection into either the deltoid or gluteal muscle.
  * Gemcitabine will be given intravenously at a dose of 600 mg/m2 over 90 minutes on Days 1 and 8 of each cycle. Docetaxel will be given intravenously at a dose of 60 mg/m2 over 60 minutes on Day 8 of each cycle. Patients started on gemcitabine at a dose of 900 mg/m2 or 750 mg/m2 or docetaxel at a dose of 75 mg/m2 per previous protocol version will be allowed to continue at that dose level
  * After Cycle 8, patients may continue on ADI-PEG 20 alone (without gemcitabine and docetaxel) upon request.
  * Treatment may continue for up to 34 cycles (103 weeks)
Arm/Group | Cohort 1, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 1, 750 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 1, 900 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel | Cohort 2, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel
All-Cause Mortality (participants affected / at risk) | 19/33 | 15/25 | 19/24 | 12/15
Serious Adverse Events (participants affected / at risk) | 14/33 | 8/25 | 13/24 | 5/15
Other Adverse Events (participants affected / at risk) | 33/33 | 25/25 | 24/24 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel (N=33) | Cohort 1, 750 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel (N=25) | Cohort 1, 900 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel (N=24) | Cohort 2, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel (N=15)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0
Mitral Valve Disease (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colonic Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper GI Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — with melena
Death NOS (General disorders) | 0 | 0 | 0 | 1
Fever (General disorders) | 1 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0
Hepatic Hemorrhage (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 1 | 1 | 2 | 1
Other (Infections and infestations) | 1 | 0 | 0 | 0 — Influenza A
Other (Infections and infestations) | 0 | 0 | 0 | 1 — COVID-19
Sepsis (Infections and infestations) | 0 | 3 | 4 | 1
Skin Infection (Infections and infestations) | 1 | 0 | 2 | 1
Upper Respiratory Infection (Infections and infestations) | 2 | 0 | 0 | 0
Other (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — Ileal Bleed due to tumor invasion
Postoperative Hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Leukemia Secondary to Oncology Chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 — Due to previous Doxorubicin
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1 — Facial
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0 | 1 | 0
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — due to disease progression
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Thromboembolic Event (Vascular disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel (N=33) | Cohort 1, 750 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel (N=25) | Cohort 1, 900 mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel (N=24) | Cohort 2, 600mg/m2 Gemcitabine Dose Level: ADI-PEG 20 + Gemcitabine + Docetaxel (N=15)
Anemia (Blood and lymphatic system disorders) | 29 | 19 | 23 | 13
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Chest Pain - Cardiac (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 2 | 2 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 2 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Blurred Vision (Eye disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 1 | 0
Retinal Tear (Eye disorders) | 0 | 1 | 0 | 0
Watering Eyes (Eye disorders) | 1 | 2 | 2 | 0
Abdominal Distention (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 1 | 3 | 1
Anal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal Mucositis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colonic Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 8 | 5 | 8 | 2
Dental Caries (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 10 | 8 | 9 | 2
Dry Mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 3 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Fecal Incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Lip Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mucositis Oral (Gastrointestinal disorders) | 6 | 5 | 3 | 2
Nausea (Gastrointestinal disorders) | 13 | 8 | 14 | 2
Oral Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Other (Gastrointestinal disorders) | 1 | 1 | 1 | 0 — Hematochezia, Generalized GI Bleed
Other (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Tooth Extraction
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 4 | 3 | 4
Chills (General disorders) | 0 | 1 | 0 | 0
Edema Face (General disorders) | 0 | 1 | 0 | 0
Edema Limbs (General disorders) | 10 | 6 | 11 | 2
Edema Trunk (General disorders) | 0 | 1 | 1 | 0
Facial Pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 23 | 22 | 18 | 5
Fever (General disorders) | 4 | 9 | 5 | 1
Flu-Like Symptoms (General disorders) | 1 | 1 | 1 | 0
Generalized Edema (General disorders) | 5 | 0 | 0 | 0
Infusion Related Reaction (General disorders) | 1 | 0 | 0 | 1
Injection Site Reaction (General disorders) | 3 | 3 | 1 | 1
Localized Edema (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 1 | 1 | 1
Other (General disorders) | 0 | 2 | 0 | 0 — Pain at Injection Site
Pain (General disorders) | 0 | 0 | 0 | 1
Allergic Reaction (Immune system disorders) | 4 | 0 | 0 | 0
Autoimmune Disorder (Immune system disorders) | 0 | 1 | 0 | 0 — Celiac Disease
Bladder Infection (Infections and infestations) | 0 | 0 | 1 | 0
Bronchial Infection (Infections and infestations) | 1 | 0 | 1 | 0
Enterocolitis Infection (Infections and infestations) | 1 | 1 | 1 | 0
Eye Infection (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Gum Infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 2 | 1 | 0 | 0
Papulopustular Rash (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0
Pleural Infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 2 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 1 | 0
Thrush (Infections and infestations) | 3 | 1 | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 5 | 4 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 3 | 5 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Other (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 — Twisted Knee, Ankle Sprain, Port Site Bleed
Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2 | 2 | 5 | 0
Alanine Aminotransferase Increased (Investigations) | 14 | 14 | 11 | 4
Alkaline Phosphatase Increased (Investigations) | 13 | 12 | 13 | 6
Aspartate Aminotransferase Increased (Investigations) | 1 | 8 | 10 | 2
Blood Bilirubin Increased (Investigations) | 2 | 6 | 7 | 2
Blood Lactate Dehydrogenase Increased (Investigations) | 2 | 0 | 1 | 0
Cardiac Troponin I Increased (Investigations) | 1 | 2 | 1 | 0
Cardiac Troponin T Increased (Investigations) | 0 | 0 | 1 | 0
Creatinine Increased (Investigations) | 7 | 5 | 9 | 1
Electrocardiogram QT Corrected Interval Prolonged (Investigations) | 1 | 1 | 0 | 0
GGT Increased (Investigations) | 0 | 0 | 0 | 1
INR Increased (Investigations) | 4 | 4 | 12 | 0
Lipase Increased (Investigations) | 0 | 0 | 2 | 0
Lymphocyte Count Decreased (Investigations) | 24 | 18 | 24 | 10
Neutrophil Count Decreased (Investigations) | 25 | 19 | 17 | 10
Other (Investigations) | 0 | 0 | 0 | 1 — Ammonia Levels Increased
Platelet Count Decreased (Investigations) | 28 | 23 | 21 | 11
Weight Loss (Investigations) | 0 | 3 | 0 | 2
White Blood Cell Decreased (Investigations) | 25 | 22 | 20 | 11
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 6 | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 5 | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 5 | 7 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 8 | 5 | 10 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 | 8 | 15 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 15 | 7 | 12 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 7 | 7 | 10 | 3
Hyponatremia (Metabolism and nutrition disorders) | 14 | 7 | 12 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 4 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 4 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 6 | 2 | 0 | 0
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 2 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Other (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 1 — Muscle "tightness", left hand pain, R axillary pain, R neck stiffness, R flank pain, "frozen thumb", hip pain
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0 — Palpable Lump RUE, Skin Pailloma R Hallux, Tumor Progression, Vaginal Cyst
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 3 | 0 | 2
Concentration Impairment (Nervous system disorders) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 5 | 2 | 0
Dysgeusia (Nervous system disorders) | 8 | 5 | 8 | 0
Extrapyramidal Disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 5 | 3 | 1
Neuralgia (Nervous system disorders) | 1 | 1 | 2 | 0
Other (Nervous system disorders) | 0 | 2 | 0 | 0 — Cerebral Hemorrhage, Plantar Sensitivity
Paresthesia (Nervous system disorders) | 2 | 2 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 9 | 5 | 10 | 0
Phantom Pain (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 2 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 2 | 0 | 0
Confusion (Psychiatric disorders) | 3 | 2 | 0 | 1
Depression (Psychiatric disorders) | 5 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 3 | 2 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 2 | 0 | 0
Hematuria (Renal and urinary disorders) | 9 | 3 | 8 | 0
Proteinuria (Renal and urinary disorders) | 7 | 7 | 7 | 0
Renal Calculi (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary Frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Genital Edema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Other (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 — Groin Pain
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 — Spotting
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 5 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 | 5 | 6 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 3 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Chest Pressure with Exertion
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Nail Changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 0
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail Loss (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Other (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 1 — Rash NOS, Nail Bed Pain, Feet Peeling, petechial rash
Palmar-Plantar Erythrodysethesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 4
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Other (Surgical and medical procedures) | 2 | 0 | 0 | 0 — minor gum transplant
Hot Flashes (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 3 | 2 | 0
Hypotension (Vascular disorders) | 1 | 4 | 3 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 0 | 0
Other (Vascular disorders) | 0 | 1 | 0 | 0 — Peripheral Edema
Thromboembolic Event (Vascular disorders) | 0 | 3 | 1 | 0 — Deep Vein Thrombosis, Pulmonary Embolism

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT03449901/Prot_SAP_002.pdf
  • Informed Consent Form (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT03449901/ICF_000.pdf